CLINICAL TRIAL: NCT02012088
Title: Phase II, Randomised, Multicentre Study With Two Treatment Arms (R-COMP Versus R-CHOP) in Newly Diagnosed Elderly Patients (≥60 Years) With Non-localised Diffuse Large B-cell Lymphoma (DLBCL)/Follicular Lymphoma Grade IIIb.
Brief Title: Clinical Trial to Evaluate R-COMP Versus R-CHOP in Newly Diagnosed Patients With Non-localised Diffuse Large B-cell Lymphoma (DLBCL)/Follicular Lymphoma Grade IIIb
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEL-R-COMP-2013
Record Dates: First submitted 2013-11-11; First posted 2013-12-16 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma
Keywords: Follicular lymphoma, large B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Doxorubicin; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RCOMP (Experimental): R-COMP Regimen:
  Day 1: Rituximab 375 mg/m2; Myocet® 50 mg/m2; cyclophosphamide 750 mg/m2; vincristine 1.4 mg/m2 (maximum 2 mg); prednisone 60 mg/m2 Days 2-5: Prednisone, 60 mg/m2 Administered every 21 days × 6 cycles
  Interventions: Drug: RCOMP
- RCHOP (Active Comparator): R-CHOP Regimen:
  Day 1: Rituximab 375 mg/m2; Doxorubicin 50 mg/m2; cyclophosphamide 750 mg/m2; vincristine 1.4 mg/m2 (maximum 2 mg); prednisone 60 mg/m2 Days 2-5: Prednisone, 60 mg/m2 Administered every 21 days × 6 cycles
  Interventions: Drug: RCHOP

INTERVENTIONS:
Drug: RCOMP — Day 1: Rituximab 375 mg/m2; Myocet® 50 mg/m2; cyclophosphamide 750 mg/m2; vincristine 1.4 mg/m2 (maximum 2 mg); prednisone 60 mg/m2 Days 2-5: Prednisone, 60 mg/m2 Administered every 21 days × 6 cycles
  Other Names: Rituximab; Myocet; Cyclophosphamide; Vincristine; Prednisone
  Arms: RCOMP
Drug: RCHOP — Day 1: Rituximab 375 mg/m2; Doxorubicin 50 mg/m2; cyclophosphamide 750 mg/m2; vincristine 1.4 mg/m2 (maximum 2 mg); prednisone 60 mg/m2 Days 2-5: Prednisone, 60 mg/m2 Administered every 21 days × 6 cycles
  Other Names: Rituximab; Doxorubicin; Cyclophosphamide; Vincristine; Prednisone 60 mg/m2
  Arms: RCHOP

SUMMARY:
The Phase II study proposed here assesses the hypothesis that replacing doxorubicin by Myocet® in the R-CHOP regimen would yield comparable antitumour efficacy with a lower cardiotoxicity for first-line treatment in elderly patients with non-localised DLBCL/Follicular lymphoma grade IIIb

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common histological subtype of non-Hodgkin's lymphoma (NHL). This is an aggressive lymphoma, with an incidence in Western countries estimated at 5-6 cases/100,000 inhabitants/year that increases with age.

Treatment for patients with DLBCL is currently based on immunochemotherapy, of which the R-CHOP regimen, which includes cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) in combination with the anti-CD20 monoclonal antibody rituximab and is administered every 21 days for a total of 6-8 cycles, is the most commonly used.

Cardiotoxicity is one of the undesirable effects that limit the use of anthracyclines, such as doxorubicin, as part of the CHOP regimen, which is caused by the formation of complexes between ferric ions and the anthracycline within the myocyte. Because of their oxidative properties, these complexes are toxic and produce highly reactive free radicals that damage the lipid membrane and lead to the cell death of myocytes. Several studies have linked the onset of cardiotoxicity with old age, high cumulative doses of doxorubicin, cardiovascular risk factors and previous heart disease, among others. Anthracycline-induced cardiotoxicity is cumulative and irreversible. Moreover, left ventricular dysfunction is an important late effect in patients with aggressive NHL who survive long term and, according to some studies, have received doxorubicin at doses higher than 200 mg/m². Cardiotoxicity may be silent or subclinical, which is usually detected as a decrease in left ventricular ejection fraction (LVEF), or clinical, with varying degrees of congestive heart failure (CHF). Depending on the symptoms, cardiotoxicity also differs between acute, subacute, late or chronic. The first is manifested at an early stage, usually as arrhythmia, transient ECG changes or pericarditis, among others, is usually reversible, is not detrimental to the continuation of treatment and is not associated with subacute and late toxicity.

Chronic cardiotoxicity could be early or late. Early-onset cardiotoxicity occurs within 1 year after anthracycline treatment and late-onset cardiotoxicity occurs more than 1 year after completion of anthracycline treatment. In the latter two, cardiotoxicity is associated with the lesion of cardiomyocytes and is therefore considered irreversible. The incidence of cardiotoxicity varies among different studies, depending on patient follow-up or the definition of cardiotoxicity used (acute, subacute or late).

In addition to clinical findings, the determination of LVEF or, more recently, the use of biomarkers, are the most commonly used methods to diagnose and assess cardiotoxicity. Regarding the identification of biomarkers, troponin I and N-terminal fragment of pro-brain natriuretic peptide (NT-proBNP) are the most commonly used and investigated in the context of clinical studies. The advantages of using biomarkers include their minimally invasive identification, which is less expensive than echocardiography, and, unlike radionuclide ventriculography, they avoid irradiation of the patient. Furthermore, the interpretation of their results does not depend on the observer's experience, thus avoiding interobserver variability. Several studies have shown the role of troponins as indicators of early anthracycline-induced cardiotoxicity or other chemotherapeutic agents, which are able to predict impaired ventricular function and higher incidence of cardiac events in patients with elevated values of this marker compared with patients with normal troponin values. Regarding the use of brain natriuretic peptides such as NT-proBNP, several studies have shown a correlation between persistently high values of this biomarker and impaired heart function parameters, in particular LVEF.

Myocet® (non-pegylated liposomal doxorubicin) is one of the several strategies developed to reduce cardiotoxicity and maintain the therapeutic efficacy of the R-CHOP regimen. Non-pegylated liposomal doxorubicin has shown a similar efficacy and less cardiotoxicity than conventional doxorubicin in the treatment of women with metastatic breast cancer. In addition, several studies in patients with NHL have shown similar response rates with regimens containing non-pegylated liposomal doxorubicin to those obtained in historical controls with conventional doxorubicin, with a low incidence of clinical and subclinical cardiovascular events. The treatment is relatively well tolerated, while myelosuppression is its most important toxicity.

Most of these phase I and II studies (with or without rituximab), which assessed Myocet® in combination with cyclophosphamide; vincristine and prednisone, showed that it is an active treatment in newly diagnosed patients with aggressive NHL.

100% of the data registered on CRFs will be source data verified. eCRDs will be used in order to register the data. Nine monitoring visits per site will be performed.

First monitoring vistit will be performed when the first patient is included Second monitoring visit willb be performed when the third patient is included Third monitoring visit will be perforemd when the fifth patient is included Fourth monitoring visit will be performed then the last patient finish study treatment One monitoring visit per year will be performed during follow-up phase.

CRO (Dynamic) Standard Operating Procedures will be used to manage the clinical trial.

Sample size of the study is based on the hypothesis of a LEVF decrease <55% in the 15% of patients assigned to R-CHOP treatment group and 5% of patients assigned to R-COMP treatment group.

Categorical variables were show by absolute and relative frequencies, including the confidence interval of 95%.

For the description of the continuous variables will be use the mean, standard deviation, median, mode, minimum and maximum, including the total number of valid values.

In the case of compare subgroups of patients, will be use for quantitative variables parametric tests or nonparametric as characteristics of the variables under study. For qualitative variables will be use Chi-square test.

Statistical analysis was planned with the SAS statistical package version 9.1 or later.

Two interim analysis will be performed when the last patient peforms the end of treatment visit and when the last patient performd the 24 months follow-up visit.

Final analysis will be performed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age
* Histological confirmed DLBCL/follicular lymphoma grade IIIb by WHO classification, with any IPI (International Prognostic Index)
* Newly diagnosed, with no previous treatment
* Non-localised stage, i.e. lymphoma that does not fit into a single radiotherapy field (including clinical stage IA with large tumour mass until stage IV) with at least one measurable lesion
* ECOG performance status 0 to 2
* Present appropriate haematologic, liver (ALT or AST < 2.5 ULN ? upper limit of normal) and renal functions (creatinine < 2.5 ULN) , unless changes are secondary to lymphoma
* LVEF at rest ? 55%, with no documented history of congestive heart failure (CHF), serious arrhythmia or acute myocardial infarction

Exclusion Criteria:

* Clinical stage I without large tumour mass or clinical stage IIA with fewer than three affected areas (stage-IIB patients are considered suitable, regardless of the number of affected areas)
* CNS infiltration
* Transformed lymphoma, although with no previous treatment, as well as other histological subtypes such as mantle cell lymphoma, peripheral T-cell lymphoma and its variants and post-transplant lymphoproliferative syndrome
* Clinically significant secondary cardiovascular disease
* Signs of any severe, acute or chronic and active infection
* Concurrent malignancy or history of other neoplasia except basal cell carcinoma (BCC) and cervical or breast carcinoma in situ (CIN)
* Patients with positive results in the HBV, HIV or HCV RNA tests
* Any previous treatment for DLBCL/follicular lymphoma grade IIIb

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Subclinical cardiac toxicity | Day 135
  Subclinical cardiac toxicity determined by the percentage of measurings experiencing a decrease in LEVF determined by echocardiography with final LEVF <55% at day 135
Subclinical cardiac toxicity | Day 225
  Subclinical cardiac toxicity determined by the percentage of measurings experiencing a decrease in LEVF determined by echocardiography with final LEVF <55% at day 225

SECONDARY OUTCOMES:
Survival | 2 and 5 years
  Event free survial, progression free survival and overall survival at 2 and 5 years.
Response rate | Day 135
  Overall response rates and complete responses evaluated by the International Harmonization Project for response criteria in lymphoma
Cardiac/cardiovascular toxicity | During 5 years
  Rate of cardiac/cardiovascular toxicity according to the CTC criteria (version 4.0) of the National Cancer Institute (NCI) during the treatment and during 5 years
Toxicity (except cardiac) | During 2 years
  No cardiotoxicity according to the CTC criteria (version 4.0) of the NCI during 24 months
Cardiac biomarkers | During 12 months
  Cardiotoxicity determined by elevated values of troponin and NT-proBNP and decreased values of LEVF determined during 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alejandro Martin, Principal Investigator — University of Salamanca; Dr. Juan Manuel Sancho, Principal Investigator — Germans Trias i Pujol Hospital; Dr. Francisco Gual, Principal Investigator — Germans Trias i Pujol Hospital
Locations (14):
- Spain (14):
  - Hospital Universitario de Alava, Vitoria-Gasteiz, Alava
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital de Cabueñes, Gijón, Asturas
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Result] Rigacci L, Mappa S, Nassi L, Alterini R, Carrai V, Bernardi F, Bosi A. Liposome-encapsulated doxorubicin in combination with cyclophosphamide, vincristine, prednisone and rituximab in patients with lymphoma and concurrent cardiac diseases or pre-treated with anthracyclines. Hematol Oncol. 2007 Dec;25(4):198-203. doi: 10.1002/hon.827. PMID 17654614
- [Result] Luminari S, Montanini A, Caballero D, Bologna S, Notter M, Dyer MJS, Chiappella A, Briones J, Petrini M, Barbato A, Kayitalire L, Federico M. Nonpegylated liposomal doxorubicin (MyocetTM) combination (R-COMP) chemotherapy in elderly patients with diffuse large B-cell lymphoma (DLBCL): results from the phase II EUR018 trial. Ann Oncol. 2010 Jul;21(7):1492-1499. doi: 10.1093/annonc/mdp544. Epub 2009 Dec 11. PMID 20007997
- [Result] Levine AM, Tulpule A, Espina B, Sherrod A, Boswell WD, Lieberman RD, Nathwani BN, Welles L. Liposome-encapsulated doxorubicin in combination with standard agents (cyclophosphamide, vincristine, prednisone) in patients with newly diagnosed AIDS-related non-Hodgkin's lymphoma: results of therapy and correlates of response. J Clin Oncol. 2004 Jul 1;22(13):2662-70. doi: 10.1200/JCO.2004.10.093. PMID 15226333
- [Result] Cardinale D, Sandri MT, Colombo A, Colombo N, Boeri M, Lamantia G, Civelli M, Peccatori F, Martinelli G, Fiorentini C, Cipolla CM. Prognostic value of troponin I in cardiac risk stratification of cancer patients undergoing high-dose chemotherapy. Circulation. 2004 Jun 8;109(22):2749-54. doi: 10.1161/01.CIR.0000130926.51766.CC. Epub 2004 May 17. PMID 15148277
- [Result] Cardinale D, Sandri MT. Role of biomarkers in chemotherapy-induced cardiotoxicity. Prog Cardiovasc Dis. 2010 Sep-Oct;53(2):121-9. doi: 10.1016/j.pcad.2010.04.002. PMID 20728699
- [Result] Cardinale D, Salvatici M, Sandri MT. Role of biomarkers in cardioncology. Clin Chem Lab Med. 2011 Sep 6;49(12):1937-48. doi: 10.1515/CCLM.2011.692. PMID 21892906
- [Derived] Sancho JM, Fernandez-Alvarez R, Gual-Capllonch F, Gonzalez-Garcia E, Grande C, Gutierrez N, Penarrubia MJ, Batlle-Lopez A, Gonzalez-Barca E, Guinea JM, Gimeno E, Penalver FJ, Fuertes M, Bastos M, Hernandez-Rivas JA, Moraleda JM, Garcia O, Sorigue M, Martin A. R-COMP versus R-CHOP as first-line therapy for diffuse large B-cell lymphoma in patients >/=60 years: Results of a randomized phase 2 study from the Spanish GELTAMO group. Cancer Med. 2021 Feb;10(4):1314-1326. doi: 10.1002/cam4.3730. Epub 2021 Jan 25. PMID 33492774
- See also: Sponsor web page — http://www.geltamo.com/